CLINICAL TRIAL: NCT00257010
Title: Long-Term, Open-Label Safety Study of Oral Almotriptan Malate 12.5 mg in the Treatment of Migraine in Adolescents
Brief Title: A 1-year Study in Adolescents to Assess the Long-term Safety of Almotriptan Malate When Treating Their Migraine Headaches
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Ortho LLC (Industry)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002827; CAPSS-368 (Other: Janssen-Ortho LLC)
Record Dates: First submitted 2005-11-18; First posted 2005-11-22 (Estimated); Results first posted 2013-12-06 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-01

CONDITIONS: Migraine
Keywords: Migraine; Almotriptan Malate; Headache; Triptan
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — almotriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Almotriptan Malate (Experimental): Patients will take one 12.5 mg almotriptan malate tablet by mouth after the onset of migraine headache pain
  Interventions: Drug: Almotriptan Malate

INTERVENTIONS:
Drug: Almotriptan Malate — Patients will take one 12.5 mg almotriptan malate tablet by mouth after the onset of migraine headache pain

SUMMARY:
The purpose of this study is to evaluate the long-term safety of almotriptan malate (a migraine headache medication) in the treatment of migraine headaches in adolescents for up to one year.

DETAILED DESCRIPTION:
Almotriptan malate, and several other treatments for migraine headaches, known as triptans, are approved for the treatment of migraine headaches in adults. To date, none of these have been approved by the Food and Drug Administration (FDA) for use in adolescents. This is an open-label, multi-center study that will enroll approximately 450 patients aged 12 - 17 years old with a history of one to 14 migraines per month for the 6 months prior to entering the study. The total study duration will be up to one year. There is a screening phase to determine if the patient is eligible for study entry, followed by an open-label treatment phase that can last up to one year. Almotriptan malate 12.5 mg tablets will be used to treat all migraine headaches during the study, as needed. The primary outcome of the study is an assessment of the long-term safety of almotriptan malate in adolescent migraine sufferers. The study hypothesis is that the almotriptan malate will be safe and well tolerated in the treatment of adolescent migraine headaches. Safety measurements will be performed at set time points during the study and will include laboratory tests, physical and neurological exams, electrocardiograms (ECGs) and the incidence of adverse events. A diary will be completed by the patient for each migraine headache for which they take almotriptan malate. Migraine pain information and almotriptan malate use will be recorded in the headache diary. An equal number of patients in the 12 - 14 year old range as the 15 - 17 year old range will be enrolled. Patients will take one 12.5 mg almotriptan malate tablet by mouth after the onset of migraine headache pain. The dose may be repeated once if the pain continues 2 hours after the first dose, but no more than 2 doses can be taken within a 24-hour period. Study medication will be taken for up to one year.

ELIGIBILITY:
Inclusion Criteria:

* Have a history of migraine for at least one year
* Have an average of 1 - 14 migraines per month for the 6 months prior to study entry
* Able to swallow oral medication
* Able to complete a headache diary
* Only taking one migraine preventive medication and on the same dose of that medication for at least 30 days before entering the study)

Exclusion Criteria:

* Have an allergy to almotriptan malate or have stopped taking almotriptan malate due to side effects
* Have 15 or more days within a month in which you have a headache
* Usually experience migraine aura (most common symptoms being visual disturbances or tingling sensations before migraine pain begins) without a headache
* Experience more than 6 non-migraine headaches per month

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 447 (Actual)
Dates: Start 2005-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Ortho LLC Clinical Trial, Study Director — Janssen-Ortho LLC
Locations (49):
- United States (49):
  - Mobile, Alabama
  - Montgomery, Alabama
  - Oxford, Alabama
  - Mesa, Arizona
  - Phoenix, Arizona
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Santa Monica, California
  - Centennial, Colorado
  - Denver, Colorado
  - Loxahatchee Groves, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Snellville, Georgia
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Des Moines, Iowa
  - Topeka, Kansas
  - Witchita, Kansas
  - Louisville, Kentucky
  - Ann Arbor, Michigan
  - Columbia, Missouri
  - Springfield, Missouri
  - St Louis, Missouri
  - Endwell, New York
  - Mineola, New York
  - Mount Vernon, New York
  - Plainview, New York
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Alcoa, Tennessee
  - Bristol, Tennessee
  - Germantown, Tennessee
  - Morristown, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - San Antonio, Texas
  - San Marcos, Texas
  - Salt Lake City, Utah
  - Madison, Wisconsin

REFERENCES:
- See also: Long-Term, Open-Label Safety Study of Oral Almotriptan Malate 12.5 mg in the Treatment ofMigraine in Adolescents — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=290&filename=CR002827_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 55 sites in the United States.
Pre-assignment Details: Of the 447 participants enrolled, 420 participants took at least one dose of study drug according to the Headache Record and were included in the analysis.
Groups:
- Almotriptan Malate: Participants received 12.5 mg almotriptan malate tablet by mouth after the onset of migraine headache pain.
Period: Overall Study
Arm/Group | Almotriptan Malate
Started | 447
Completed | 319
Not Completed | 128
Not completed — Lack of Efficacy | 11
Not completed — Lost to Follow-up | 53
Not completed — Withdrawal by Subject | 34
Not completed — Adverse Event | 10
Not completed — various | 11
Not completed — no headache reported | 9

BASELINE CHARACTERISTICS:
Arm/Group | Almotriptan Malate
Number analyzed (Participants) | 447
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.4 (1.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 245
  Male | 202

OUTCOME MEASURES:

1. Primary Outcome: Number of Pain Free Headaches at 2 and 24 Hours Post-Dose
Description: Headache pain free is defined as a decrease in baseline pain intensity from severe, moderate or mild to no pain, without the use of supplemental pain medication and/or anti-emetic medication (including a second dose of study medication) within 2 (or 24) hours of first dose of study medication. Sustained pain free is defined as pain free at 2 and 24 hours without the use of supplemental pain medication and/or anti-emetic medication (including a second dose of study medication) within 24 hours.
Time Frame: 2 hours and 24 hours post-dose
Population: Intent-to-Treat (ITT) population is defined as all enrolled participants who took at least one dose of study medication and for whom at least one post-dose efficacy assessment was available.
Measure: Number; unit: Number of headaches
Units Other Than Participants: headaches
Arm/Group | Almotriptan Malate
Number analyzed (Participants) | 420
Number analyzed (headaches) | 7941
Number of headaches
  Headaches Pain Free at 2 hours | 3218
  Headaches Pain Free at 24 hours | 5236
  Headaches Sustained Pain Free at 24 hours | 3048

2. Secondary Outcome: Number of Headaches Achieving Pain Relief at 2 and 24 Hours Post-Dose
Description: Headache pain relief is defined as a decrease in baseline pain intensity from either severe or moderate intensity to mild or no pain, without the use of supplemental pain medication and/or anti-emetic medication (including a second dose of study medication) within 2 (or 24) hours of first dose of study medication. Sustained pain relief is defined as pain relief at 2 and 24 hours without the use of supplemental pain medication and/or anti-emetic medication (including a second dose of study medication) within 24 hours.
Time Frame: 2 hours and 24 hours post-dose
Population: as for outcome 1
Measure: Number; unit: Number of headaches
Units Other Than Participants: headaches
Arm/Group | Almotriptan Malate
Number analyzed (Participants) | 420
Number analyzed (headaches) | 6099
Number of headaches
  Headaches Pain Relief at 2 hours | 3765
  Headaches Pain Relief at 24 hours | 4182
  Headaches Sustained Pain Relief at 24 hours | 3384

3. Secondary Outcome: Number of Headaches With Photophobia
Description: Occurrence and intensity of photophobia post-dose of study medication. Photophobia is an abnormal sensitivity to or intolerance of light, especially by the eyes.
Time Frame: Baseline (after onset of migraine headache pain and before treatment), 2 hours and 24 hours post-dose
Population: as for outcome 1
Measure: Number; unit: Number of headaches with photophobia
Units Other Than Participants: headaches
Arm/Group | Almotriptan Malate
Number analyzed (Participants) | 420
Number analyzed (headaches) | 8052
Number of headaches with photophobia
  At baseline | 6164
  At 2 hours | 3150
  At 24 hours | 936

4. Secondary Outcome: Number of Headaches With Phonophobia
Description: Occurrence and intensity of phonophobia post-dose of study medication. Phonophobia is an abnormal sensitivity to or intolerance of noise.
Time Frame: Baseline (after onset of migraine headache pain and before treatment), 2 hours and 24 hours post-dose
Population: as for outcome 1
Measure: Number; unit: Number of headaches with phonophobia
Units Other Than Participants: headaches
Arm/Group | Almotriptan Malate
Number analyzed (Participants) | 420
Number analyzed (headaches) | 8052
Number of headaches with phonophobia
  At baseline | 5783
  At 2 hours | 2847
  At 24 hours | 805

5. Secondary Outcome: Number of Headaches With Nausea
Description: Occurrence and intensity of nausea post-dose of study medication. Nausea is a feeling of sickness characterized by gastrointestinal distress and an urge to vomit.
Time Frame: Baseline (after onset of migraine headache pain and before treatment), 2 hours and 24 hours post-dose
Population: as for outcome 1
Measure: Number; unit: Number of headaches with nausea
Units Other Than Participants: headaches
Arm/Group | Almotriptan Malate
Number analyzed (Participants) | 420
Number analyzed (headaches) | 8052
Number of headaches with nausea
  At baseline | 3262
  At 2 hours | 1785
  At 24 hours | 542

6. Secondary Outcome: Number of Headaches With Vomiting
Description: Occurrence and intensity of vomiting post-dose of study medication. Vomiting is an act or instance of disgorging the contents of the stomach through the mouth also called emesis.
Time Frame: Baseline (after onset of migraine headache pain and before treatment), 2 hours and 24 hours post-dose
Population: as for outcome 1
Measure: Number; unit: Number of headaches with vomiting
Units Other Than Participants: headaches
Arm/Group | Almotriptan Malate
Number analyzed (Participants) | 420
Number analyzed (headaches) | 8052
Number of headaches with vomiting
  At baseline | 357
  At 2 hours | 258
  At 24 hours | 107

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Almotriptan Malate
Serious Adverse Events (participants affected / at risk) | 8/420
Other Adverse Events (participants affected / at risk) | 282/420
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Almotriptan Malate (N=420)
Bradycardia Foetal (Cardiac disorders) | 1
Intussusception (Gastrointestinal disorders) | 1
Appendicitis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Gun Shot Wound (Injury, poisoning and procedural complications) | 1
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1
Major Depression (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Almotriptan Malate (N=420)
Anaemia (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Tachycardia (Cardiac disorders) | 1
Ventricular Hypertrophy (Cardiac disorders) | 1
Cerumen Impaction (Ear and labyrinth disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 2
Motion Sickness (Ear and labyrinth disorders) | 1
Eye Allergy (Eye disorders) | 1
Eye Irritation (Eye disorders) | 1
Hypermetropia (Eye disorders) | 1
Myopia (Eye disorders) | 1
Scotoma (Eye disorders) | 1
Vision Blurred (Eye disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 10
Aphthous Stomatitis (Gastrointestinal disorders) | 1
Chapped Lips (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 8
Dry Mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 1
Food Poisoning (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 3
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 5
Gingival Swelling (Gastrointestinal disorders) | 1
Hypoaesthesia Oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 25
Salivary Gland Disorder (Gastrointestinal disorders) | 1
Stomach Discomfort (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 1
Tooth Disorder (Gastrointestinal disorders) | 1
Tooth Impacted (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 23
Chills (General disorders) | 2
Fatigue (General disorders) | 3
Influenza Like Illness (General disorders) | 2
Malaise (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Oedema Peripheral (General disorders) | 1
Pain (General disorders) | 5
Pyrexia (General disorders) | 15
Vessel Puncture Site Bruise (General disorders) | 1
Biliary Colic (Hepatobiliary disorders) | 1
Biliary Dyskinesia (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Drug Hypersensitivity (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 6
Seasonal Allergy (Immune system disorders) | 1
Abscess Limb (Infections and infestations) | 1
Acute Sinusitis (Infections and infestations) | 2
Acute Tonsillitis (Infections and infestations) | 1
Bacterial Infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 9
Bronchitis Acute (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Coccidioidomycosis (Infections and infestations) | 1
Conjunctivitis Infective (Infections and infestations) | 2
Ear Infection (Infections and infestations) | 8
Eye Infection (Infections and infestations) | 2
Gastritis Viral (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Gastroenteritis Viral (Infections and infestations) | 15
Gonorrhoea (Infections and infestations) | 1
Gynaecological Chlamydia Infection (Infections and infestations) | 1
Herpes Simplex (Infections and infestations) | 2
Herpes Zoster (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 2
Infectious Mononucleosis (Infections and infestations) | 3
Influenza (Infections and infestations) | 14
Localised Infection (Infections and infestations) | 1
Mastitis (Infections and infestations) | 1
Nail Infection (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 52
Otitis Externa (Infections and infestations) | 4
Otitis Media (Infections and infestations) | 5
Pelvic Inflammatory Disease (Infections and infestations) | 1
Pertussis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 11
Pharyngitis Streptococcal (Infections and infestations) | 18
Pneumonia (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Respiratory Tract Infection (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 29
Skin Infection (Infections and infestations) | 1
Staphylococcal Infection (Infections and infestations) | 1
Subcutaneous Abscess (Infections and infestations) | 1
Tinea Infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 3
Upper Respiratory Tract Infection (Infections and infestations) | 28
Urinary Tract Infection (Infections and infestations) | 5
Vaginal Candidiasis (Infections and infestations) | 1
Varicella (Infections and infestations) | 2
Viraemia (Infections and infestations) | 1
Viral Infection (Infections and infestations) | 13
Viral Rhinitis (Infections and infestations) | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 8
Vulvovaginal Mycotic Infection (Infections and infestations) | 1
Vulvovaginitis Trichomonal (Infections and infestations) | 1
Animal Bite (Injury, poisoning and procedural complications) | 1
Chemical Eye Injury (Injury, poisoning and procedural complications) | 1
Clavicle Fracture (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 7
Contusion (Injury, poisoning and procedural complications) | 6
Epicondylitis (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 2
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Foot Fracture (Injury, poisoning and procedural complications) | 1
Forearm Fracture (Injury, poisoning and procedural complications) | 1
Foreign Body Trauma (Injury, poisoning and procedural complications) | 1
Gun Shot Wound (Injury, poisoning and procedural complications) | 1
Hand Fracture (Injury, poisoning and procedural complications) | 3
Head Injury (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Joint Injury (Injury, poisoning and procedural complications) | 2
Joint Sprain (Injury, poisoning and procedural complications) | 12
Ligament Injury (Injury, poisoning and procedural complications) | 3
Ligament Sprain (Injury, poisoning and procedural complications) | 1
Limb Injury (Injury, poisoning and procedural complications) | 4
Medical Device Pain (Injury, poisoning and procedural complications) | 2
Muscle Strain (Injury, poisoning and procedural complications) | 2
Periorbital Haematoma (Injury, poisoning and procedural complications) | 1
Post-Traumatic Pain (Injury, poisoning and procedural complications) | 2
Procedural Pain (Injury, poisoning and procedural complications) | 3
Skin Laceration (Injury, poisoning and procedural complications) | 1
Thermal Burn (Injury, poisoning and procedural complications) | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 3
Alanine Aminotransferase Increased (Investigations) | 1
Aspartate Aminotransferase Increased (Investigations) | 1
Blood Glucose Increased (Investigations) | 2
Blood Triglycerides Increased (Investigations) | 1
Blood Urine Present (Investigations) | 1
Electrocardiogram Pr Prolongation (Investigations) | 1
Electrocardiogram QRS Complex Prolonged (Investigations) | 1
Epstein-Barr Virus Test Positive (Investigations) | 1
Glucose Urine Present (Investigations) | 1
Haematocrit Decreased (Investigations) | 1
Haemoglobin Decreased (Investigations) | 1
Lymph Nodes Scan Abnormal (Investigations) | 1
Neutrophil Count Increased (Investigations) | 1
Protein Urine (Investigations) | 2
Protein Urine Present (Investigations) | 2
Red Blood Cell Count Decreased (Investigations) | 1
Red Blood Cells Urine (Investigations) | 1
Spleen Palpable (Investigations) | 1
Weight Decreased (Investigations) | 2
Weight Increased (Investigations) | 2
White Blood Cell Count Increased (Investigations) | 1
White Blood Cells Urine Positive (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Increased Appetite (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 6
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 5
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 3
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4
Scoliosis (Musculoskeletal and connective tissue disorders) | 1
Temporomandibular Joint Syndrome (Musculoskeletal and connective tissue disorders) | 2
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Disturbance in Attention (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 8
Facial Neuralgia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 8
Hyperreflexia (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 2
Loss of Consciousness (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 6
Paraesthesia (Nervous system disorders) | 2
Paraesthesia Oral (Nervous system disorders) | 1
Post-Traumatic Headache (Nervous system disorders) | 2
Psychomotor Hyperactivity (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 6
Syncope (Nervous system disorders) | 5
Tension Headache (Nervous system disorders) | 1
Affective Disorder (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Attention Deficit/Hyperactivity Disorder (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 8
Mood Altered (Psychiatric disorders) | 1
Sleep Disorder (Psychiatric disorders) | 1
Stress (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Enuresis (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 7
Menstruation Irregular (Reproductive system and breast disorders) | 2
Oligomenorrhoea (Reproductive system and breast disorders) | 1
Ovarian Cyst Ruptured (Reproductive system and breast disorders) | 1
Allergic Cough (Respiratory, thoracic and mediastinal disorders) | 1
Allergic Respiratory Symptom (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Asthma Exercise Induced (Respiratory, thoracic and mediastinal disorders) | 3
Bronchial Hyperactivity (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 17
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 27
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 4
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 5
Acne (Skin and subcutaneous tissue disorders) | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 6
Drug Eruption (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 2
Hirsutism (Skin and subcutaneous tissue disorders) | 1
Pain of Skin (Skin and subcutaneous tissue disorders) | 2
Petechiae (Skin and subcutaneous tissue disorders) | 2
Pigmentation Disorder (Skin and subcutaneous tissue disorders) | 1
Precancerous Skin Lesion (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 5
Rash Generalised (Skin and subcutaneous tissue disorders) | 1
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1
Scar (Skin and subcutaneous tissue disorders) | 1
Skin Striae (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Vitiligo (Skin and subcutaneous tissue disorders) | 1
Tooth Extraction (Surgical and medical procedures) | 1
Hot Flush (Vascular disorders) | 1
Systolic Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days